CLINICAL TRIAL: NCT05756244
Title: A Prospective Cohort Study Evaluating Peripartum Anticoagulation Management Among Pregnant Women With Venous Thromboembolism and Its Impact on Patient Outcomes
Brief Title: PRospective Evaluation of Peripartum Anticoagulation ManaGement for ThrOmboembolism
Acronym: PREP and GO
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB21-0795
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy Related; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PREP and GO study is an international multicentre prospective cohort evaluating anticoagulation management strategies around labor and delivery and the postpartum period.

DETAILED DESCRIPTION:
The goal of this study is to provide quality data using standardized outcome definitions on postpartum bleeding events, venous thromboembolism (VTE) risk, delivery experience outcomes and health care utilization for intrapartum and postpartum anticoagulation management among pregnant individuals on low-molecular-weight heparin (LMWH) for prevention of treatment of VTE.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Requires anticoagulation during the antepartum period of pregnancy for a VTE indication, including at least one of:

  1. Objectively confirmed VTE (DVT, superficial vein thrombosis [SVT], PE or unusual site thrombosis) diagnosed during the current pregnancy;
  2. Objectively confirmed VTE diagnosed in a prior pregnancy;
  3. Objectively confirmed VTE diagnosed when not pregnant;
  4. Inherited or acquired thrombophilia requiring anticoagulation.
* Receiving any dose or type of LMWH during the antepartum period

Exclusion Criteria:

* Anticoagulation for a non-VTE indication, including prosthetic heart valves, atrial fibrillation, prevention of placenta-mediated pregnancy complications, or prevention of recurrent pregnancy loss (participants can be included with a diagnosis of antiphospholipid syndrome (APS) with or without thrombotic events)
* Unable to provide or declined consent.
* Home or birthing centre planned delivery.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant individuals on anticoagulation for VTE-related indications
Sampling Method: Non-Probability Sample
Enrollment: 825 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of MB and CRNMB | Delivery up to 6 weeks postpartum
  To estimate the combined incidence of major bleeding (MB) and clinically relevant non-major bleeding (CRNMB) for the six most common antepartum strategies.

SECONDARY OUTCOMES:
Practice Patterns | Prior to delivery and following delivery
  To determine the practice patterns of intrapartum and postpartum anticoagulant management for pregnant individuals on LMWH for VTE indications across participating centres.
MB and CRNMB incidence in the immediate and 6 W postpartum period | Within 24 hours of delivery and up to 6 weeks postpartum
  To estimate the incidence of MB and CRNMB in the immediate postpartum period (within 24 hours) and up to 6 weeks postpartum for each antepartum strategy.
MB and CRNMB incidence up to 6 W postpartum related to anticoagulation resumption | 6 weeks postpartum
  To estimate the incidence of MB and CRNMB up to 6 weeks postpartum, based on the time and dose of postpartum anticoagulation resumption.
Incidence of VTE | Delivery to 6 weeks postpartum
  To estimate the incidence of symptomatic objectively confirmed VTE up to 6 weeks postpartum for each antepartum strategy.
Wound Hematoma | Delivery to 6 weeks postpartum
  To estimate the incidence of wound hematoma complications up to 6 weeks postpartum for each antepartum strategy.
Anti-Xa levels | Delivery
  To compare anti-Xa levels on admission for delivery in individuals with and without immediate postpartum MB and CRNMB.
Hemoglobin Levels around Delivery | Before and after delivery
  To compare a change in hemoglobin levels before and after delivery in individuals with and without immediate postpartum MB and CRNMB.
Patient Experience | Delivery
  To describe delivery experience outcomes including neuraxial anesthesia (eligible vs. preferred vs. actual), patient satisfaction, and patient choice relating to delivery management options.
Healthcare Utilization | Before and after delivery
  To quantify healthcare utilization including hospital length of stay, postpartum length of stay, repeat procedures and induction of labor resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Skeith, MD, Principal Investigator — University of Calgary; Isabelle Malhamé, MD, Principal Investigator — McGill University; Kinga Malinowski, MD, Principal Investigator — University of Toronto
Locations (14):
- Duke University Hospital, Durham, North Carolina, United States
- Canada (10):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - BC Women's Hospital and Health Centre, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - McMaster University Medical Centre, Hamilton, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Montfort Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - The Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- Aarhus University Hospital, Aarhus, Denmark
- Le Centre Hospitalier Universitaire of Saint-Etienne, Saint-Etienne, France
- Hopitaux universitaires de Geneve, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Please contact study PI for requests.